CLINICAL TRIAL: NCT02977923
Title: Decreasing REcurrent Pain and Anxiety in Medical Procedures With a Pediatric Population: a Pilot Study
Acronym: DREAM-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Quebec Nursing Intervention Research Network (Other)
Responsible Party: Principal Investigator, Sylvie Le May, RN, PhD, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1383
Record Dates: First submitted 2016-11-26; First posted 2016-11-30 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Pain; Anxiety; Burns; Child; Injuries
Keywords: Virtual reality; Immersive distraction; Oculus rift; Virtual world; Virtual environment; Procedural pain; Procedural anxiety; Acute pain; Pain management; Anxiety; Children, Child; Kid, Kids; Pediatric, Pediatrics; Young children; Burns; Burn injuries; Burn unit; Physiotherapy; Physical therapy; Burn dressing; Dressing change; Non-pharmacological, nonpharmacological; Clinical Research; Nursing Practice; Trauma
MeSH Terms: conditions — Pain; Anxiety Disorders; Burns; Wounds and Injuries; Pain, Procedural; Acute Pain; Agnosia; Deafness, Autosomal Recessive 1A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pharmacological treatment (Active Comparator): According to the unit's protocol and adjusted to each participant's age, weight and condition by the anesthetist and pain clinic nurse.
  Interventions: Other: Standard pharmacological treatment
- VR distraction via Oculus Rift (Experimental): In addition to standard pharmacological treatment, Virtual reality distraction through the use of Oculus Rift® will be used as the experimental intervention. The Oculus Rift (Consumer version) is made of two Oled panels with a resolution of 1200p running at 90Hz. It has very effective 360 degree positional tracking and integrated 3D audio. These combine to produce a high level of immersion, with high photorealism while maintaining the low latency necessary to induce presence and prevent cybersickness. The child, depending on the site of the injury, will have the opportunity to interact with the game. Video games, approved by healthcare professionals with extensive experience in pediatrics, were adapted for children and tailored to minimize cyber sickness.
  Interventions: Device: VR distraction via Oculus Rift

INTERVENTIONS:
Device: VR distraction via Oculus Rift — In addition to standard pharmacological treatment, Virtual reality distraction through the use of Oculus Rift® will be used as the experimental intervention. The Oculus Rift (Consumer version) is made of two Oled panels with a resolution of 1200p running at 90Hz. It has very effective 360 degree positional tracking and integrated 3D audio. These combine to produce a high level of immersion, with high photorealism while maintaining the low latency necessary to induce presence and prevent cybersickness. The child, depending on the site of the injury, will have the opportunity to interact with the game. Video games, approved by healthcare professionals with extensive experience in pediatrics, were adapted for children and tailored to minimize cyber sickness.
  Arms: VR distraction via Oculus Rift
Other: Standard pharmacological treatment — according to the unit's protocol and adjusted to each participant's age, weight and condition by the anesthetist and pain clinic nurse.
  Arms: Standard pharmacological treatment

SUMMARY:
Children with injuries, including burns, experience severe pain intensity during medical procedures despite the increasing doses of analgesics. Current guidelines on pediatric procedural pain management recommend the combination of non-pharmacological and pharmacological interventions to enhance pain management and decrease the numerous side effects of analgesics. Virtual reality (VR) has gained growing consideration as a non-pharmacological method as it engages multiple senses and allows interactions with a virtual world. Oculus Rift ® (OR) is a new technology in VR that provides more immersiveness, at a relatively low cost, and could probably improve the management of pain and anxiety in wound care.

Overall hypothesis: Distraction by VR via the OR, in combination with the standard pharmacological treatment, is a feasible, acceptable and satisfactory method for the management of pain and anxiety during wound-related treatments in children with injuries.

Note that this pilot study will precede a larger trial aimed at assessing the effect of virtual reality distraction via the Oculus Rift ® (DREAM-T: NCT02947243)

DETAILED DESCRIPTION:
BACKGROUND:

Injuries, including burns, are the leading cause of morbidity and mortality in children. They are associated with a lot of pain that is difficult to treat and can impede recovery, cause high levels of anxiety and alter future pain behaviors, resulting, at times, in chronic pain, paresthesia, or depression. Pain can also decrease participation in treatments such as physiotherapy resulting in poor health outcomes. Beyond the immediate pain experience, children may also develop pain memory circuits. Procedural pain is still largely managed pharmacologically mostly through the use of opioids, benzodiazepines, and other pharmacological agents which cause a lot of side effects and do not always provide sufficient pain reduction. In recent years, the effectiveness of multimodal approaches combining medication with non-pharmacological interventions for procedural pain relief has been highlighte. Distraction techniques engaging multiple senses may grab the child's attention more than the techniques that only engage one sense (e.g, music), hence, the increasing interest in more immersive and interactive methods of distraction such as Virtual Reality (VR).

VR is an active distraction method that allows the user to interact with an immersive environment generated by a computer stimulating different senses. A review of studies on VR, mostly conducted with adult burn patients, showed a 35 to 50% reduction in procedural pain while using VR. However, despite promising results, the use of VR in healthcare settings has been limited, mainly due to its high cost. Reviews have highlighted the need for more research but mostly for the development of more portable, less expensive and more developed VR systems that would promote pain reduction during burn procedures especially for children with burn injuries who are considered one of the most challenging burn populations. However, there has been a breakthrough in technology since 2014 when big scale companies started investing in VR development for commercial gaming. Facebook purchased the Oculus Rift (OR) for mass production allowing access to the latest technology in VR at a relatively low cost. OR is a VR tool that provides a wide field of view (FOV), high-resolution display, integrated 3D audio and motion detection. In addition, it's highly immersive properties could help achieve more analgesia compared to other VR techniques as a review has shown that the sense of presence influences the effectiveness of VR-based analgesia. The sense of presence is a subjective psychological state of consciousness of being in the virtual world whereas immersiveness refers to the physical environment that could be quantified by measuring the field of view or the peripheral vision in the VR goggles. The availability of inexpensive yet highly immersive VR goggles such as OR could increase the use of VR in pain management and burn settings while significantly improving its cost-effectiveness. A single case study assessed the feasibility of a VR intervention via OR in one child of 11 years old with burn injuries during occupational therapy. The study showed a reduction in pain intensity and pain unpleasantness experienced by the patient, without any side effects. To our knowledge, no other studies have tested the feasibility of OR for procedural pain management in children with injuries undergoing painful physiotherapy treatments or wound care.

AIM: The aim of this pilot clinical trial is to assess the acceptability and feasibility of VR distraction using the OR in children with injuries undergoing wound-related treatments (physiotherapy or dressing change). We also plan to evaluate the feasibility of the design and to predict appropriate sample size for a larger-scale clinical trial.

METHODS:

Design: Within-subject/crossover study design. Each child will serve as his own control and will receive both standard and experimental treatment during the same treatment session through a randomized order.

Sample and Setting: Convenience sampling on the surgical-trauma unit at CHU Ste-Justine, of children presenting with an injury.

Interventions. A) Standard pharmacological treatment as per the unit's protocol. B) VR distraction through the use of OR.The video games were developed by our team with a personalized care content tailored to the children's developmental stage and to maximize the feeling of immersion and minimize cybersickness, and approved by a team of healthcare professionals in pediatric care.

Study proceedings: Physiotherapy sessions and dressing changes typically last between 20 to 30 minutes. The duration will be divided into two sequences of the same duration (10 to 15 minutes) where the participant receives the same care by the same healthcare professional. For one sequence, only the standard treatment will be administered and for the other sequence, patients will receive the standard treatment in addition to VR via OR in a randomized order.

Measures: Pain and anxiety measures will be taken before the treatment session at (T1), after the first sequence of the session (T2) and after the second sequence of the session (T3) followed by a measure of nurses' satisfaction level via a questionnaire developed and pretested by the team. We will collect data on the average doses of analgesics administered before and during the session, and the side effects experienced in addition to the design's feasibility outcomes: participants recruited each month, adherence to study protocol.

Data analysis: Quantitative analysis. Mean differences in pain scores between sequences will be compared using Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

* suffer from a burn or another injury requiring wound dressing change or physiotherapy
* presence of a consenting parent who can understand, read and write either French or English

Exclusion Criteria:

* Requiring intensive care
* Having a diagnosed cognitive impairment
* Are unconscious or intubated during dressing change or physiotherapy sessions
* Suffering from epilepsy (considering the nature of the intervention)
* Allergic to opioids or other analgesics used for standard pharmacological treatment
* Having injuries on the face preventing the use of the Oculus Rift helmet

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Acceptability | T4, immediately after the procedure completion, before leaving the procedure room
  To assess the acceptability including the satisfaction of healthcare professionals regarding the use of the VR distraction via Oculus Rift during the treatment session. Pre-tested tailored questionnaire including satisfaction and acceptability outcomes (tolerance, positive and negative aspects, secondary effects).

SECONDARY OUTCOMES:
Mean Pain Score | T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session
  Numerical Rating Scale (NRS) ranging from 0 to 10; 0=no pain to 10=pain as bad as it could be
Pain Experience | T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  Graphic Rating Scale (GRS) consisting of seven items to measure the cognitive, the affective and the sensory components of pain
Expected Anxiety | Baseline (T1)
  Children's Fear Scale (CFS)
Experienced Anxiety | T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  Children's Fear Scale (CFS)
Comfort Level | T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  Behavioural observation scale of comfort level for child burn victims (OCCEB-BECCO)
Pain Memory | 24 hours after the procedure (T5)
  A measure of the child's memory of pain using the same measure (NRS) administered during the initial data collection to assess this construct
Anxiety Memory | 24 hours after the procedure (T5)
  A measure of the child's memory of anxiety using the same measure (CFS) administered during the initial data collection to assess this construct
Range Of Motion | Baseline (T1); T2: 10 minutes within the session (immediately after the first sequence of the session); T3: 20 minutes within the session (immediately after the second sequence of the session)
  (only for physiotherapy sessions) Using a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, RN, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Ste. Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No